CLINICAL TRIAL: NCT01428336
Title: The Value of 25 mcg Cortrosyn Stimulation Test to Assess Adult HPA Axis
Brief Title: Value of 25 mcg Cortrosyn Stimulation Test
Acronym: 25CST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1945
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Intervention Model Description: Every participant underwent the four interventional tests in random sequence
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Active Comparator): Subjects will undergo three ACTH stimulation test using a dose of 1 ug cotrosyn, 25 ug cortrosyn, 250ug cortrosyn and one Insulin tolerance test
  Interventions: Procedure: 1 ug ACTH stimulation test; Procedure: 250 ug ACTH stimulation test; Procedure: 25 ug Cortrosyn stimulation test; Procedure: Insulin tolerance test
- Volunteers (Active Comparator): Subjects will undergo three ACTH stimulation test using a dose of 1 ug cotrosyn, 25 ug cortrosyn, 250ug cortrosyn and one Insulin tolerance test
  Interventions: Procedure: 1 ug ACTH stimulation test; Procedure: 250 ug ACTH stimulation test; Procedure: 25 ug Cortrosyn stimulation test; Procedure: Insulin tolerance test

INTERVENTIONS:
Procedure: 1 ug ACTH stimulation test — 1 ug cortrosyn dose
Procedure: 250 ug ACTH stimulation test — ACTH stimulation test will be done using 250 ug cortrosyn dose
Procedure: 25 ug Cortrosyn stimulation test — ACTH stimulation test using a 25 ug cortrosyn dose
Procedure: Insulin tolerance test — subjects will undergo an insulin tolerance test

SUMMARY:
The diagnosis of secondary AI is vital to prevent catastrophic events in patients. An optimal test should have a very low margin of error with high sensitivity and specificity, be easy and safe to administer, and have distinct cut off values. Both 1 ug and 250 ug doses have their limitations. Based on our experience over the past six years, we hypothesize that 25 ug ACTH stimulation test may eliminate some of the shortcomings of the LDST (1 ug) and SDST (250 ug). This is supported by our preliminary data and the study by Oelkers et al, which looked at ACTH levels following various doses of cortrosyn injections.

Therefore we propose a head to head comparison of 25 ug, 250 ug and 1 ug dose using ITT as gold standard.

DETAILED DESCRIPTION:
The study consisted of two groups of adult patients 18 to 65 years of age. The first group (G1, n=10) included patients with hypothalamic/pituitary disease with at least one pituitary axis deficiency other than ACTH deficiency. The patients had the following diagnoses: acromegaly (n=1), prolactinoma (n=2), non-secreting pituitary macroadenomas (n=3), pituitary cholesterol granuloma (1), uncharacterized pituitary stalk lesion(1),recurrent null cell adenoma(1) and craniopharyngioma (n=1). The second group (G2, n=12) comprised healthy volunteers. The three CSTs and ITT were done in random order and separated by a median of 22 days (range, 2 - 64 days) from each other. Cortisol levels were measured at 30 and 60 minute (min) during CSTs. A peak cortisol cut-off of 18 μg/dl was used as the pass criterion during ITT. The result of total cortisol levels during ITT were used to determine free cortisol cut-offs during CSTs and ITT. None of the patients had pituitary surgery within six weeks prior to enrollment and none of the women were on estrogen.

Patients in G1 had to be on at least 3 months of stable hormone replacement for hormone deficiencies. All control subjects (G2) had normal TSH, free T4 and prolactin levels. All premenopausal women in the control group had a history of regular, age appropriate menses and none took birth control pills within 3 months of study entry. Postmenopausal subjects had appropriately elevated FSH concentration. All men in the control group had normal FSH and total testosterone levels.

Exclusion criteria included: inability of subject to give an informed consent, pregnancy, patients with diabetes mellitus type 1 and type 2, any pituitary insult such as pituitary surgery in the past 6 weeks, elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3 times the upper limit of normal, renal failure (defined as serum creatinine more than 2 mg/dl), history of malignancy in the last 5 years, severe acute illness and patients on opioid (fentanyl, oxycodone, hydrocodone, acetaminophen/hydrocodone) treatment. In addition, patients with a history of coronary artery disease, cerebrovascular disease, congestive heart failure, arrhythmias, or seizure disorder, were excluded due to the potential risk during ITT.

Study procedures: Patients with HPA axis disorders and control subjects interested in the study were contacted by the research team for a screening interview. A complete medical history was obtained for each study participant. For female participants, a reproductive history was taken. All women in reproductive age group had a negative urine pregnancy test.

All study participants were instructed to fast overnight for 12 hours prior to testing. Six patients were on glucocorticoid replacement and were instructed to hold their medication for 24 hours prior to their dynamic testing. All the tests were conducted at the Clinical Research Unit on site at the Cleveland Clinic. The study was approved by the Cleveland Clinic Institutional Review Board. All subjects signed an informed consent.

Cosyntropin Stimulation tests: The 250 µg cosyntropin vial was reconstituted with 1 ml of 0.9% saline and used the same day. 25 µg cosyntropin was prepared by reconstituting the 250 µg vial with 1 ml of 0.9% saline and withdrawing 0.1 ml for each injection. The unused reconstituted cosyntropin vials were discarded at the end of the day. 1 µg cosyntropin was prepared by diluting the 250 µg in 250ml of 0.9% saline and withdrawing 1ml for intravenous injection. Reconstituted solution for 1 µg dose was refrigerated and used for up to a month. During the CSTs, sFC and TC levels were drawn at baseline (t=0 min) and then at 30 and 60 min after 1µg (IV), 25 µg (IM) and 250µg (IM) cosyntropin doses.

ITT: The test was initiated between 0800 and 0900 hrs, after an overnight fast. Regular human insulin 0.10 - 0.15 units /kg was administered intravenously, with target blood glucose less than 40 mg/dL. Additional insulin bolus was administered, if needed, to achieve the target glucose value. Administration of oral or intravenous dextrose was allowed if the subject developed signs of symptomatic hypoglycemia. Blood glucose levels were checked at 0, 15, 30, 45, 60, 90 and 120 min and sFc and TC were drawn at 0, 30, 45, 60, 90 and 120 min.

Assays: The screening labs for control subjects TSH, free T4, prolactin and complete metabolic profile and bedside blood glucose tests were done at the Cleveland Clinic lab. The screening labs for FSH, Testosterone, and samples of TC and sFC were analyzed at Quest Diagnostics Nichols Institute, San Juan Capistrano, CA 92675, USA.

TC was measured using Liquid Chromatography Mass Spectrometry (LCMS). The intra assay coefficient of variation (CV) were 3.0-4.6% at 15.9 and 202.7 µg /dl, respectively. The inter-assay CV were 4.8 and 7.6% at 15.2 and 189.9 µg /dl, respectively. sFC was measured using LCMS after separating bound and unbound cortisol by equilibrium dialysis. The intra assay CVs were 7.4 and 9.3 % at 0.36 and 2.17 µg /dl, respectively. The inter-assay CVs were 9.4 and 9.8% at 0.36 and 2.17 µg/dl, respectively.

Statistical analysis: Patient groups were compared on categorical factors using Pearson chi-square tests and Fisher exact tests. Continuous measures were evaluated using Wilcoxon rank sum tests. Sensitivity(SE) and specificity(SP) for each of the CSTs were estimated using optimal cut-offs from ROC curves, with respect to ITT as the gold standard. Youden's Index, which identifies the largest combination of SE and SP for each test was used to identify the optimal cut-off for each test. Tests were compared on SE and SP using McNemar's test. Pearson's correlation coefficient was used to measure the strength of association of peak cortisol levels among pairs of testing methods. Ninety-five percent confidence intervals were produced for all the correlation, SE, and SP estimates. Comparisons of the correlations were performed using the methods by Meng, Rosenthal, and Rubin (1992) to compare the correlations and calculate 95% confidence intervals for the difference among the tests [17]. Lower bounds of these intervals above a zero value was considered statistically significant evidence that the 25-µg test is a better test, while lower bounds at least as high as -0.15 was used to determine non-inferiority at those respective margins. Analyses were performed using R software (version 3.1; Vienna, Austria) and SAS software (version .3; Cary, NC).

ELIGIBILITY:
Inclusion Criteria:

* hypothalamic-pituitary-adrenal disorders

Exclusion Criteria:

* under 18 or older than 65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seenia Peechakara, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Department of Endocrinology, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients | Volunteers
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Every participant underwent three ACTH stimulation test using a dose of 1 ug cotrosyn, 25 ug cortrosyn, 250ug cortrosyn and one Insulin tolerance test
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Volunteers | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pearson Correlation of the Total Cortisol Levels Between the ITT and CSTs
Description: Correlation of total cortisol levels of 1 ug, 25 ug and 250 ug cortrosyn stimulation test with Insulin Tolerance test is described in the outcome table
Time Frame: 1 hour for the CST interventions and 2 hour for the ITT interventions
Population: Correlation of total cortisol levels with 1 ug, 25 ug and 250 ug cortrosyn stimulation test with Insulin Tolerance test is described in the outcome table. The two groups of patients and volunteers were combined to get a full range of values for each intervention.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- Patients + Volunteers: Every participant underwent three ACTH stimulation test and one Insulin tolerance test.
Arm/Group | Patients + Volunteers
Number analyzed (Participants) | 22
correlation coefficient
  Peak 1 ug ACTH stimulation test | 0.8 [0.57 to 0.91]
  Peak 25 ug ACTH stimultion test | 0.86 [0.69 to 0.94]
  60-minute 250ug ACTH stimulation test | 0.93 [0.83 to 0.97]
  30-minute 250ug ACTH stimulation test | 0.92 [0.82 to 0.97]
Statistical Analysis 1: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. Peak 1ug CST correlation with ITT; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = 0.06, 95% CI 2-sided [-0.20 to 0.60]
Statistical Analysis 2: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. Peak 250ug CST correlation with ITT; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = -0.07, 95% CI 2-sided [-0.69 to -0.01]
Statistical Analysis 3: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. 30-minute 250ug CST correlation with ITT; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = -0.06, 95% CI 2-sided [-0.65 to 0.04]

2. Secondary Outcome: Pearson Correlation of Free Cortisol Values During CSTs With ITT
Description: Correlation of free cortisol levels of 1 ug, 25 ug and 250 ug cortrosyn stimulation test with Insulin Tolerance test is described in the outcome table
Time Frame: 1 hour for the CST interventions and 2 hour for the ITT interventions
Population: Correlation of free cortisol levels with 1 ug, 25 ug and 250 ug cortrosyn stimulation test with Insulin Tolerance test is described in the outcome table. The two groups of patients and volunteers were combined to get a full range of values for each intervention.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Patients + Volunteers
Number analyzed (Participants) | 22
correlation coefficient
  Peak 1ug ACTH stimulation test | 0.58 [0.20 to 0.80]
  Peak 25ug ACTH stimulation test | 0.70 [0.39 to 0.87]
  60- minute 250ug ACTH stimulation test | 0.88 [0.74 to 0.95]
  30-minute 250ug ACTH stimulation test | 0.89 [0.74 to 0.95]
Statistical Analysis 1: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. Peak 1ug CST correlation with ITT - free cortisol; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = 0.12, 95% CI 2-sided [-0.24 to 0.65]
Statistical Analysis 2: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. Peak 250ug CST correlation with ITT - free cortisol; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = -0.18, 95% CI 2-sided [-0.91 to -0.15]
Statistical Analysis 3: Comparison: Patients + Volunteers; Analysis comparing Peak 25ug CST correlation with ITT vs. 30-minute 250ug CST correlation with ITT - free cortisol; Test type: Non-Inferiority — A non-inferiority region of 0.15 for the difference in correlations is expected; Difference in correlation = -0.19, 95% CI 2-sided [-0.94 to -0.14]

3. Secondary Outcome: Peak Total Cortisol Values
Description: Peak total cortisol values during cortrosyn stimulation tests(CST)
Time Frame: 1 hour for the CST interventions and 2 hour for the ITT interventions
Measure: Median (Full Range); unit: ug/dl
Arm/Group | Patients | Volunteers
Number analyzed (Participants) | 10 | 12
ug/dl
  Insulin Tolerance Test | 23.3 [20.2 to 25.9] | 16.6 [1.1 to 26.1]
  1 ug ACTH stimulation test | 23.4 [16.7 to 31.9] | 14.5 [2.2 to 28.4]
  25 ug ACTH stimulation test | 22.0 [16.4 to 28.6] | 17.4 [2.0 to 24.9]
  30 min 250 ug ACTH stimulation test | 22.3 [18.8 to 27.8] | 16.1 [1.8 to 25.8]
  60 min 250 ug ACTH simulation test | 25.0 [21.9 to 31.5] | 19.1 [2.4 to 29.4]

ADVERSE EVENTS:
Groups:
- 1ug Cortrosyn Dose Stimulation Test: Subjects will undergo an ACTH stimulation test using a dose of 1 ug cotrosyn
  ACTH stimulation test: 1 ug cortrosyn dose
  1 ug cortrosyn test: Subjects will undergo an ACTH test using a 1 ug dose cortrosyn
- 250 ug Cortrosyn Dose Stimulation Test: Subjects will undergo an ACTH stimulation test using 250 ug cortrosyn dose
  250 ug ACTH stimulation test: ACTH stimulation test will be done using 250 ug cortrosyn dose
- 25 ug Cortrosyn Stimulation Test: Subjects will undergo an ACTH stimulation test using a 25 ug cortosyn dose
  25 ug Cortrosyn stimulation test: ACTH stimulation test using a 25 ug cortrosyn dose
Arm/Group | 1ug Cortrosyn Dose Stimulation Test | 250 ug Cortrosyn Dose Stimulation Test | 25 ug Cortrosyn Stimulation Test | Insulin Tolerance Test
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
Small number of participants Cortisol Binding globulin was not measured

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No